CLINICAL TRIAL: NCT01229969
Title: A Pilot Study of the Wii Fit as a Low-Cost Virtual Reality System to Evaluate Balance Ability in Older Adults
Acronym: WiiFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Theodore Johnson II, M.D., M.P.H., Site Director, Birmingham/Atlanta VA GRECC, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-060390
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Falls, Accidental
Keywords: falls, balance problems, gaming systems, balance assessments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeuroCom EquiTest® System (Experimental): Measure balance assessment (test for Sensory Organization Test (SOT) and Limit of Stability (LOS).
  Interventions: Other: NeuroCom EquiTest® System
- Wii Fit (Experimental): Determine if the Wii Fit is valid and feasible in detecting balance problems in older adults
  Interventions: Other: Wii Fit Balance Games

INTERVENTIONS:
Other: Wii Fit Balance Games — Ski Slaloms and Table Tilt
  Other Names: Ski Slaloms and Table Tilt
  Arms: Wii Fit
Other: NeuroCom EquiTest® System — Sensory Organization Test (SOT) and Limit of Stability (LOS).
  Other Names: SOT and LOS
  Arms: NeuroCom EquiTest® System

SUMMARY:
Accidental falls in older adults are highly prevalent and a major source of morbidity. Over 30% of people aged 65 or older fall each year with about half of these cases being recurrent. Falls may result in head trauma, bone fractures, and even death and are leading cause of both nonfatal and fatal injuries in older adults. The Nintendo Wii Fit is a suite of exercise and fitness video games using a balance board periphery developed for the Wii console. The purpose of this study is to determine the feasibility and validity of the Nintendo Wii Fit, in detecting balance problems in older community dwelling adults.20 ambulatory older adults will be recruited to participate in this study.Subject will be asked to complete 1 study visit. In this visit information will be gathered about the subjects overall health including fall assessments. Qualified subjects will be randomized into two study groups where one group will begin the study with Wii Fit testing followed by NeuroCom EquiTest evaluation and the other group in reversed order.

DETAILED DESCRIPTION:
Accidental falls in older adults are highly prevalent and a major source of morbidity. Over 30% of people aged 65 or older fall each year with about half of these cases being recurrent. Falls may result in head trauma, bone fractures, and even death and are leading cause of both nonfatal and fatal injuries in older adults. Falls are also costly. An estimate $20 billion dollars annually has been spent on hip fractures associated with falls; this amount is projected to rise in the next decade. Risk factors for falls in the elderly are usually multi-factorial. These include increasing age, environmental factors, acute or chronic illness, medication use, cognitive impairment, sensory deficits, and balance and gait impairment.

The Nintendo Wii Fit system is engaging, low-cost, and standardized and may be a feasible exercise modality to improve balance in the elderly. While virtual reality use in a research context is not new, few studies of commercially available low-cost video games with virtual reality capabilities have been done. These have demonstrated encouraging results, indicating a potential use for rehabilitation in both children and adults.

Twenty ambulatory older individuals age 60 and older who reside in the community will be recruited to participate in this study.This group of participants will be selected to represent the general community dwelling older adults as much as possible. They will demonstrate a wide range of ability in terms of their balance and mobility in which some are healthy (non-fallers), some with risks of falling, and some fallers. Efforts will be made to have equal distribution among these three groups.

Subjects will be consented for the research study and we will ask questions about age, gender, educational background, medical history, and any falls in past year. They will also be evaluated clinically before the actual study to assess vision, cognitive status, and balance.

Qualified subjects will be randomized into two study groups where one group will begin the study with Wii Fit testing followed by NeuroCom EquiTest evaluation and the other group in reversed order. This counterbalancing between subjects is designed to negate any potential order effect. Balance data collected from the NeuroCom EquiTest will be compared to the performance scores obtained from playing the two Wii Fit balance games to determine whether the performance scores on the two Wii Fit balance games are indicative of the participants' balance ability.All study interventions are completed in a 1 day session.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 60 years of age or older
2. Reside in the community
3. Who are with and without balance or gait issues

Exclusion Criteria:

1. Impaired mental status, patient scores <21 on Montreal Cognitive Assessment (MoCA)
2. Unable to ambulate without an assistive walking device
3. Cannot stand independently for 20 minutes of testing over a 30min period
4. Unstable medical conditions

   1. Active cardiopulmonary
   2. Degenerative neuro-sensory conditions
   3. Severe pain with weight bearing
5. Vision Impairment
6. Weighing more than 300 pounds (150kg)
7. Used Wii Fit equipment in the past

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Feasibility and validity of the Wii Fit gaming system in detect balance problems in older adults | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Theodore M Johnson, MD,MPH, Principal Investigator — Atlanta Veteran Affairs Adminstration, Emory University School of Medicine
Locations (1):
- Atlanta VA Medical Center, Atlanta, Georgia, United States